CLINICAL TRIAL: NCT05214092
Title: Cortical Contributions to Frequency-Following Response Generation and Modulation; Post-Operative Outcomes
Brief Title: Cortical Contributions to FFR: Post-Op Outcomes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Taylor Abel, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY21100033; R01DC013315 (NIH)
Record Dates: First submitted 2022-01-12; First posted 2022-01-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Language
MeSH Terms: conditions — Language

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurosurgical Patients (Experimental): Patient participants with previously excised tissue within Heschl's gyrus (as dictated by clinical care)
  Interventions: Behavioral: Speech sound stimulation

INTERVENTIONS:
Behavioral: Speech sound stimulation — Participants will listen to repetitive speech sound stimuli, presented through headphones, which will induce a neural response (frequency-following response) to be measured via electroencephalography and pupillometry

SUMMARY:
The purpose of this study is to better understand cortical contributions of the human temporal lobe to the frequency-following response. Frequency-following responses (FFR) are electrophysiological recordings that reflect phase-locked activity of neural ensembles in the auditory pathway and are used as an indicator of the integrity of supra-threshold speech processing. FFR was first studied in subcortical areas, but recent consensus in the literature supports the notion that it is an integrated response between subcortical and cortical neural populations. The proposed study aims to deconstruct the role of the cortex in generating and modulating the FFR. The research team will build a novel computational model of FFR mechanisms and use EEG recordings from participants who have undergone resection of lesions in Heschl's gyrus to validate model predictions.

DETAILED DESCRIPTION:
The purpose of this study is to better understand the cortical contribution of the human temporal lobe to the generation and modulation of frequency-following responses (FFR).

The specific aims of this study is as follows:

1. To build a novel computational model of cortical feedforward mechanisms involved in FFRs.
2. To test model predictions of cortical removal in human participants who have undergone surgical resection of Heschl's gyrus lesions.

The hypothesis to be tested for the previously listed purposes and aims are as follows:

1. When cortical areas involved in generating and modulating the FFR, in this case Heschl's gyrus, are removed or inactivated, the FFR response will be attenuated.

The frequency-following response has been used extensively in auditory processing literature as a minimally invasive method of recording the integrity of supra-threshold speech processing. It was once considered to be reflective of only subcortical activity in structures like the brainstem, however a recent consensus has been reached in research on the topic that supports the notion of cortical neural population involvement in FFR as well.

The pilot study conducted under the initial parent grant for this study (Online Modulation of Auditory Brainstem Responses to Speech) proposed that subcortical auditory processing is not a hard-wired mechanism in the human brain but is rather continuously fine-tuned to stimuli by top-down expectations. This study further demonstrated that stimulus predictability, attention, and category-relevance have a robust effect on response fidelity and can modulate the FFR. The current study proposes to study the same effects and response patterns in cortical structures. Limited studies to date have investigated the effect of auditory cortex lesions on the FFR and existing studies did not account for the variables investigated in this study that are proposed to have a significant effect on modulation of FFRs.

Even though FFR is widely accepted as a metric for measuring the integrity of speech encoding, there remains a poor understanding of the neural generators of this response. A few studies to date have already identified abnormal or dysfunctional FFR in certain clinical populations like ADHD and autism spectrum disorders. The proposed study additionally seeks to identify the potential translational utility of FFR as a biomarker for clinical conditions.

This study is innovative as data from this study will allow researchers to build a novel computational model of cortical feedforward and feedback mechanisms, which will be tested in patient participants who have undergone surgical resection of Heschl's gyrus lesions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 13-25 years old
* Undergoing medically necessary surgical resection of Heschl's gyrus lesion
* Monolingual English speakers
* Receptive and expressive language within normal limits
* Normal or corrected-to-normal visual acuity
* Normal hearing acuity in each ear (as determined during an audiometric assessment)
* Nonverbal IQ within normal limits
* No history of autism spectrum disorder or attention-deficit hyperactivity disorder

Exclusion Criteria:

* Significant medical or neuropsychological impairment that would result in the patient being unable to participate in study activities
* History of autism or ADHD

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Pitch Decoding Accuracy | During sEEG-EEG recording sessions, up to 3 hours total
  Pitch decoding accuracy will be measured as a stimulus-to-response correlation between stimulus pitch (in Hz) and scalp-recorded frequency-following responses (FFR). Hidden Markov models (HMMs) will be used to decode stimulus identity information from recorded FFRs.
Frequency-Following Response Magnitude | During sEEG-EEG recording sessions, up to 3 hours total
  The frequency-following response magnitude will be measured by analyzing the time-domain averaged spectral peak of scalp-recorded FFRs.
Cortical Phase-Locking Limits of Frequency-Following Response | During sEEG-EEG recording sessions, up to 3 hours total
  Phase-locking limits of FFRs will be measured by comparing phase coherence of stimulus waveforms and scalp-recorded FFRs. The phase-locking limit will be determined as a function of dependence on stimulus frequency.
Predictability Effects of Cortical Resection on Pitch Decoding Accuracy | During follow-up research sessions, at least 6-months post-sEEG
  The predictability effects of cortical resection on pitch decoding accuracy will be measured via comparison of decoding accuracies obtained in Outcome 1 and values predicted by a previously created computational model of frequency-following response constrained by data from neurotypical participants.
Predictability Effects of Cortical Resection on Frequency-Following Response Magnitude | During follow-up research sessions, at least 6-months post-sEEG
  The predictability effects of cortical resection on frequency-following response magnitude will be measured via comparison of response magnitude measurements obtained in Outcome 3 and values predicted by a previously created computational model of frequency-following response constrained by data from neurotypical participants.
Predictability Effects of Cortical Resection on Phase-Locking Limits of Frequency-Following Response | During follow-up research sessions, at least 6-months post-sEEG
  The predictability effects of cortical resection on phase-locking limits of the frequency-following response will be measured via comparison of phase-locking limits obtained in Outcome 3 and values predicted by a previously created computational model of frequency-following response constrained by data from neurotypical participants.

CONTACTS AND LOCATIONS:
Overall Officials: Taylor Abel, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The individual deidentified participant data intended to be shared include the individual participant data that underlie the results to be reported in published articles after deidentification.
  Other documents that will be available include the study protocol, statistical analysis plan, and analytic code.
  Data will be available as soon as possible following publication, but no later than one year upon completion. There is no end date.
  IPD will be made available for any purpose via open access.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available as soon as possible, but no later than one year upon completion of the study.
Access Criteria: Our data will be made publicly available online as soon as possible. Data will be easily and widely accessible.

REFERENCES:
- [Background] Arehart KH, Kates JM, Anderson MC. Effects of noise, nonlinear processing, and linear filtering on perceived music quality. Int J Audiol. 2011 Mar;50(3):177-90. doi: 10.3109/14992027.2010.539273. PMID 21319935
- [Background] Coffey EBJ, Nicol T, White-Schwoch T, Chandrasekaran B, Krizman J, Skoe E, Zatorre RJ, Kraus N. Evolving perspectives on the sources of the frequency-following response. Nat Commun. 2019 Nov 6;10(1):5036. doi: 10.1038/s41467-019-13003-w. PMID 31695046
- [Background] White-Schwoch T, Anderson S, Krizman J, Nicol T, Kraus N. Case studies in neuroscience: subcortical origins of the frequency-following response. J Neurophysiol. 2019 Aug 1;122(2):844-848. doi: 10.1152/jn.00112.2019. Epub 2019 Jul 3. PMID 31268800